CLINICAL TRIAL: NCT06186609
Title: Efficacy and Safety of PD-1 Inhibitor Combined With Radiotherapy in Treatment of Elderly Esophageal Squamous Cell Cancer
Brief Title: PD-1 Inhibitor Combined With Radiotherapy for Elderly ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Weiwei Yu, professor, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02121998
Record Dates: First submitted 2023-01-02; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Elderly patient; Esophageal Cancer; PD-1 inhibitor; Radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment Arm (Experimental): PD-1 inhibitor combined with radiotherapy
  Interventions: Drug: PD-1 inhibitor 200mg per three to four weeks, for one year

INTERVENTIONS:
Drug: PD-1 inhibitor 200mg per three to four weeks, for one year — PD-1 inhibitor delivered 200mg once before radiotherapy and 200mg every 3-4 weeks after radiotherapy for one year.
  Radiotherapy:56-60Gy/28-30 fraction.
  Other Names: radiotherapy

SUMMARY:
Concurrent chemoradiotherapy is now considered to be the standard treatment modality for esophageal cancer patients who are medically unfit for surgery. However, elderly patients have limitations in their ability to tolerate concurrent chemoradiotherapy in comparison to nonelderly patients because of medical comorbidities and reduced functional reserve of organs. Immune checkpoint inhibitors, including PD-1 inhibitor, have been used in a large number of clinical studies on esophageal cancer and have achieved certain results. PD-1 inhibitor combined with radiotherapy may be a new strategy for elderly patients with esophageal cancer. This study aims to explore the efficacy and safety of PD-1 inhibitor combined with radiotherapy in the treatment of elderly patients with esophageal cancer. PD-1 inhibitor was delivered 200mg once before radiotherapy and 200mg every 3-4 weeks after radiotherapy for one year.

DETAILED DESCRIPTION:
Study Design Primary Purpose: To investigate the safety and efficacy of PD-1 inhibitor combined with radiotherapy for elderly patients with esophageal squamous cell carcinoma.

Study Phase: Phase II Intervention Model: PD-1 inhibitor combined with radiotherapy Number of Arms: One Masking: No Allocation: 68 patients for one single group Enrollment: 68 patients Eligibility Criteria Inclusion Criteria: 1. ≥ 70 year-old, 2. Esophageal squamous cell carcinoma with stage II to IVA, 3. No previous surgery, radiotherapy or chemotherapy of cancer was allowed, 4. Estimated survival time ≥ 3 months, 5. KPS ≥ 70, 6. No serious diseases of important organs, 7. Signed consent forms voluntarily.

Exclusion Criteria: 1. Psychopath, 2. History of other malignant disease which has not been cured, 3. Severe autoimmune disease, 4. Joining other clinical trial prior this study.

Intervention: PD-1 inhibitor delivered 200mg once before radiotherapy and 200mg every 3-4 weeks after radiotherapy for one year. Radiotherapy:56-60Gy/28-30 fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 70 years or above
2. Treatment naive patients with pathology proven esophageal squamous cell carcinoma that was inoperable or refuse surgery and who could not tolerate concurrent chemoradiotherapy
3. Stage II-IVa according to the AJCC TNM staging system
4. Estimated survival time ≥ 3 months
5. Karnofsky performance score ≥70
6. Normal blood routine, liver and kidney function less than 2 times of the normal upper limit
7. Without mental disorders, cooperate with treatment and follow-up
8. Have fully understood this study and voluntarily signed the informed consent

Exclusion Criteria:

1. Esophageal bronchial fistula or esophageal mediastinal fistula
2. Patients who have participated in other clinical trials before this treatment
3. Severe heart, liver and/or kidney dysfunction
4. Serious infectious diseases
5. EC who has received surgery, chemotherapy,PD-1 inhibitor or radiotherapy
6. Severe autoimmune disease
7. Relapse disease or distant metastasis
8. Combined with other malignant tumors.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Two years
  The time from the start of treatment to disease progression as assessed by the treating physicians in the study (investigator-assessed)

SECONDARY OUTCOMES:
Overall Survival | Three years
  The time from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yu Weiwei, Principal Investigator — Department of Radiation Oncology, Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China